CLINICAL TRIAL: NCT04040907
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Oral Doses of XNW3009 in Healthy Adult Subject
Brief Title: The the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of XNW3009 in Health Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XNW3009-1-02
Record Dates: First submitted 2019-07-02; First posted 2019-08-01 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Intervention Model Description: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XNW3009 (Active Comparator)
  Interventions: Drug: XNW3009
- XNW3009 placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XNW3009 — XNW3009 is a small molecule hURAT1 inhibitor
  Arms: XNW3009
Drug: Placebo — Placebo and active drug will have the same appearance
  Arms: XNW3009 placebo

SUMMARY:
XNW3009 is a small molecule hURAT1 inhibitor developed independently by Sinovent Pty Ltd., and is intended to treat gout-related hyperuricemia.

Uricosuric drugs increase urinary uric acid excretion by blocking renal tubular reabsorption of urate. The human urate transporter 1( hURAT1) is responsible for the majority of the reabsorption of filtered urate, and the mutations in the hURAT1 gene have been demonstrated to be responsible for urate non-homeostasis.

This is a randomized, double-blind, placebo-controlled, dose-escalation study to investigate the safety, tolerability, PK and PD of XNW3009 after administration of single (Part A) and multiple (Part B) oral doses in healthy adult subjects. Approximately six sequential dose panels (single oral doses of 1, 5, 10, 20, 35 and 50 mg XNW3009) will be evaluated in SAD and approximately three sequential dose panels (ten consecutive days for respectively daily oral doses of 10, 20,35 mg, QD) will be evaluated in MAD.

ELIGIBILITY:
Inclusion Criteria:

1. Female (of non-child-bearing potential) or male, 18-45 years of age (both inclusive) at the time of screening;
2. Able to give signed written informed consent form, and agree to comply with protocol restrictions, including refraining from consuming alcohol, caffeinated beverages (i.e. tea, coffee, etc.), and tobacco or nicotine containing products from 24 hours before D-2 until the last PK blood sample collection is finished; Able to remain in-house for the confinement period of the study without interruption;
3. Body mass index (BMI, weight [kg]/height [m]2) within 18.0-32.0 kg/m2 (both inclusive);
4. No clinically significant abnormal values on vital signs, B ultrasound and 12-lead electrocardiogram (ECG). QT interval corrected for heart rate according to Fridericia's formula (QTcF) must be within the following ranges: QTcF ≤450 msec for male subjects, and QTcF ≤470 msec for female subjects. One repeat assessment is permitted.
5. Serum uric acid (sUA) level 4 mg/dL (0.24 mmol/L) to 8 mg/dL (0.48 mmol/L) for male and 3.5 mg/dL (0.21 mmol/L) to 8 mg/dL (0.48 mmol/L) for female during screening;
6. No clinically significant abnormal findings noted during screening for medical history and physical examination, or clinically significant abnormal results during screening clinical laboratory tests, including WBC, liver function and kidney function. One repeat assessment is permitted at the discretion of the Investigator;
7. If male and if engaging in sexual intercourse with a female partner of childbearing potential, willing to use a condom in addition to having the female partner use a highly effective method of female contraception (See Section 5.5.3.1) from the time of first study drug administration until the EOS visit. This requirement does not apply to subjects in a same sex relationship or subjects with female partners of non-childbearing potential. Male subjects must also be willing to not donate sperm for the same period.
8. If female, be of non-childbearing potential: e.g. post-menopausal for ≥12 consecutive months with follicle stimulating hormone (FSH) ≥40 mIU/mL at Screening; or surgical sterilization for at least 90 days prior to screening e.g., tubal ligation or hysterectomy. Note: Provision of documentation is not required for female sterilization, verbal confirmation is adequate.
9. Negative urine drug screen and alcohol breath testing at screening and Day-2. Note: Screening urine drug test/ alcohol breath testing may be repeated once if deemed appropriate by the investigator.

Exclusion Criteria:

* 1. Subjects who have a clinically relevant intolerance or allergy to drugs, or are known or suspected to have hypersensitivity to any ingredient in the investigational products or other URAT1 inhibitors; 2. Have a history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs. Note: a subject who has had an appendectomy or hernia repair can be enrolled in the study; 3. Subjects with a history or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urological, or psychiatric disorders; 4. Current or chronic history of liver disease or known hepatic or biliary abnormalities, including but not limited to ALT, alkaline phosphatase and bilirubin >ULN.

  5. Current or history of cardiac arrhythmias (symptomatic or asymptomatic); 6. Recent or current serious infection (within 30 days of screening). Examples include cellulitis, pneumonia, septicemia. Subjects with mild upper respiratory tract infection may be enrolled at the discretion of the investigator; 7. Estimating glomerular filtration rate (using the Modification of Diet in Renal Disease method based on serum creatinine and actual age) < 90 ml/min/1.73m2; 8. Major illness or surgery (except for minor outpatient surgery) within past 3 months of study Day 1, or planned surgery during study; 9. Subjects with intolerance to direct venipuncture; 10. Subjects with a history of, or signs and symptoms associated with, renal calculi or gout; 11. Known or suspected history of drug abuse within the past 2 years or presence of drug abuse within 3 months before screening, or evidence of such abuse on laboratory assays at screening and Day -2 unless explained by a therapeutic dose of a prescribed medication that was ceased at least 14 days prior to Day 1. Up to 1 repeat permitted; 12. Habitual use of tobacco or nicotine products or smoking within 3 months (more than 5 cigarettes per day) prior to screening, and, unwilling to refrain from use of tobacco and nicotine containing products from 24 hours before Day -2 until completion of the confinement period; 13. Unwilling to refrain from caffeinated beverages (i.e. tea, coffee, etc) from 24 hours before Day -2 until completion of the confinement period; 14. Participation in any clinical study with an investigational drug, biologic or device within 4 weeks or 5 times the half-life of the specific drug/biologics (whichever is longer), prior to dosing; 15. Donated blood >400 mL or significant blood loss equivalent to 400 mL or received blood transfusion within 3 months of screening, or donated blood >200 mL or significant blood loss equivalent to 200 mL within 1 month prior to screening; or plans to donate blood during the study; 16. Malignancy within 5 years of screening visit (excluding non-melanoma skin cancer that has been resected); 17. Recent administration or plans to receive administration of live vaccine within 12 weeks before Day 1 up to 30 days after the last dose of IP; 18. Use of any other drug, including prescription and over-the-counter medications, within 7 days prior to the first dose of study medication should be discussed with the Investigator. Where appropriate, such medication should be ceased prior to dosing. The subject may be enrolled if the medication taken or residual drug present is not expected to interfere either with subject safety or study results.
  * Paracetamol at a dose of <2 g in 24 hours but no more than 1 g in 4 hours;
  * Dietary vitamins may be allowed at the discretion of the investigator (e.g. Vitamin D taken at a standard replacement dose, and at a time remote from IP administration);
  * Herbal supplements are not permitted; 19. Use of food or beverages likely to influence liver metabolism 14 days prior to the first dose of the study drug (e.g. star fruit, pomelos, grapefruit & seville oranges); 20. History of significant alcohol abuse within 6 months of screening or any indication of regular use of more than 14 units of alcohol per week (1 Unit=360 mL of beer or 45 mL of alcohol 40% or 150 mL of wine) and, unwilling to refrain from consumption of alcohol from 24 hours before Day -2 until completion of the confinement period; 21. Positive screening test for any one or more: serum hepatitis B surface antigen (HBsAg), hepatitis C antibody, or HIV; 22. Pregnant or lactating women; 23. Subject who is considered unsuitable for participating in the study in the opinion of investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Evaluate incidence and severity of adverse eventsadministration in healthy adult subjects. | From day1 to day7 for Part A
  An AE is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.Adverse events will be coded using.
Evaluate incidence and severity of adverse eventsadministration in healthy adult subjects. | From day1 to day24for Part B
  An AE is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.Adverse events will be coded using.
Evaluate clinically significant changes from baseline in physical examinations | From day1 to day7 for Part A
  Physical examinations will be performed by a study delegated registered physician.Any findings made during the physical examination must be noted regardless of if they are part of the subject's medical history.
Evaluate clinically significant changes from baseline in physical examinations | From day1 to day24 for Part B
  Physical examinations will be performed by a study delegated registered physician.Any findings made during the physical examination must be noted regardless of if they are part of the subject's medical history.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetic of maximum plasma concentration | From day1 to day4 for Part A
  Blood samples will be collected serially for analysis throughout the study period.
Evaluate the pharmacokinetic of maximum plasma concentration | From day1 to day14 for Part B
  Blood samples will be collected serially for analysis throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Salman, Principal Investigator — Linear Clinical Research
Locations (1):
- Linear Clinical Research, Perth, West Austrialia, Australia

IPD SHARING:
Plan to Share IPD: Undecided